CLINICAL TRIAL: NCT01020929
Title: Incidence of Simultaneous Epidural and Intravascular Injection During Cervical and Lumbosacral Transforaminal Epidural Injections
Brief Title: Incidence of Simultaneous Epidural and Intravascular Injection
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: SU-09222009-3980; 16750 (Other: Stanford University)
Record Dates: First submitted 2009-11-05; First posted 2009-11-26 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Spinal Diseases
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Blunt Coude — Type of needle tip
Device: Quincke — Type of needle tip
Device: Trucath — Type of needle tip

SUMMARY:
The investigator hopes to learn the incidence of needle placement in both the epidural and intravascular space, and learn mixed epidural-intravascular pattern related to needle type, gauge, and level of injection. We also hope to evaluate the length of fluoroscopy time when using real time fluoroscopy during contrast dye injection, evaluate the radiation exposure to the hands of the physician during this protocol, and confirm the incidence fo intravascular injection and sensitivity of needle flash of blood, In the lumbar spine, vascular contrast patterns are more than twice as likely to appear simultaneous to the anticipated epidural pattern, than they are to occur alone. This is important since practitioners are more likely to miss a vascular pattern that occurs simultaneous to epidural spread, than they are to occur alone. The incidence of intravascular penetration in cervical transforaminal epidural injections is known to exceed that of lumbar injections, however no study has determined the incidence of simultaneous epidural and vascular injection in the cervical spine. This study may prove that real time fluoroscopy during contrast injection is warranted to prevent intravascular injection and resultant side effects to support this as standard of care.

Intermittent fluoroscopy can yield false-negative results for intravascular injection when simultaneous epidural and intravascular injection occurs. This could lead to an increased risk of complication from intravascular injection of medications and reduce overall efficacy. No studies to date have quantified the incidence of needle placement located in both the intravascular space and epidural space simultaneously.

DETAILED DESCRIPTION:
Any patient undergoing a lumbar or cervical transforaminal epidural, as ordered by their treating physician will provide written informed consent before the procedure is conducted. The contents of the consent forms will be used to explain the study to patients. There are no drug treatments associated with the study other than those which are part of the existing treatment plan. There is no subject randomization. Subjects will be recruited consecutively.

Patients with pregnancy, coagulopathy, systemic infection, allergy to contrast dye, mentally disabled or those whom are unable to give informed consent will be excluded from the study.

1. One experienced physician (>5 years experience) will use intermittent fluoroscopy to place needle for transforaminal epidural position using standard techniques. The physician will then use real time fluoroscopy when injecting the contrast solution to determine pattern of contrast flow (his standard of care).
2. For each individual epidural site (each level and side per patient per setting counted as separate injections) the following will be identified:

   1. Patients age
   2. Diagnosis (reason for epidural) i.e. spinal stenosis, HNP, DDD
   3. Procedure level
   4. Gauge of needle
   5. Type of needle tip
   6. Aspiration of blood in needle hub pre-injection
   7. Contrast pattern using real time fluoroscopy
   8. Number of attempts of needle positioning
   9. Total fluoro time per case
3. The physician will routinely wear a ring radiation badge to determine average radiation exposure to his hand.
4. Analyze results
5. Confirm incidence of intravascular pattern per level and determine incidence of mixed intravascular-epidural pattern per level.
6. Quantify average fluoro exposure time and compare to average flouro time of identical procedures using intermittent fluoroscopy.

All of the procedures for this protocol are standard of care.

All data is collected during the procedure. There will be no follow-ups after the procedure.

We will be asking participants if they are willing to be contacted regarding future research studies that may be of interest to them.

ELIGIBILITY:
Inclusion:

1. Any patient undergoing a lumbar or cervical transforaminal epidural, as ordered by their treating physician.
2. Ability to give informed consent.

Exclusion:

1. Pregnancy
2. Coagulopathy
3. Systemic infection
4. Allergy to contrast dye
5. Mentally disabled or those whom are unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to enroll a total of 500 subjects ( 250 subjects undergoing cervical and 250 subjects undergoing lumbosacral transforaminal epidural injection ) ;(iii) patients will have radiculopathies, herniated discs, and spinal stenosis coming to Stanford for an epidural steroid injection
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Presence or Absence of Vascular Patterns | At the time of injection

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Smuck, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States